CLINICAL TRIAL: NCT03602105
Title: Better Before - Better After: Prehabilitation Program for Older Patients Awaiting Total Hip Replacement. A Randomised Controlled Trial
Brief Title: Better Before - Better After: Prehabilitation Program for Older Patients Awaiting Total Hip Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/503
Record Dates: First submitted 2018-06-06; First posted 2018-07-26 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Arthritis of Hip
Keywords: exercise; prehabilitation; arthritis; quality of life; osteoarthritis; rehabilitation
MeSH Terms: conditions — Motor Activity; Arthritis; Osteoarthritis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Exercise interventions for 6-12 weeks. Adherence is monitored with day journals
  Interventions: Behavioral: Exercise
- Control group (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Exercise — Exercises in group and/or individually
  Arms: Intervention group

SUMMARY:
Health professions need to prepare for the large increase in the number of older people with OA requiring health services including TJA surgery. Older age and poor physical function influences the postoperative prognosis of TJA. At discharge from hospital after TJA, studies have shown that gait speed can be severely impaired among older patients.

The investigators hypothesize that an exercise program of 6-12 weeks will be beneficial for patients that are undergoing TJA.

DETAILED DESCRIPTION:
More than 300.000 Norwegians above 20 years of age have osteoarthritis (OA) . There has been a significant increase in the prevalence of OA over the decades. In the United States knee OA affects 19% of adults aged 45 years or older. OA is associated with an extensive high economic and personal burden, largely attributable to the effects of disability, comorbid disease, and the expense of treatment.

Given the aging population, the number of total joint arthroplasty procedures (TJA) for hip and knee is likely to increase substantially. In light of poor physical function prior to surgery among older patients and the likelihood of an added decrease during hospitalization and risk of poorer outcome after surgery, it is hypothesised that prehabilitation (preoperative exercise) would improve outcomes after surgery, however evidence for its efficacy is still lacking

ELIGIBILITY:
Inclusion Criteria:

* Participants 70 years or older living at home with residential address in the county of Oslo or Akershus scheduled for elective primary total hip replacement due to end-stage osteoarthritis.
* Harris Hip Score >60.
* Participants must also be capable in Norwegian and be able to follow exercise sessions.

Exclusion Criteria:

* Patients with known rheumatoid arthritis or medical contraindications or those who are scheduled for revision of hip arthroplasty
* Unable to speak and understand the Norwegian language.
* Patients with neurological disorders affecting gait
* Medical contraindications for exercise

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in gait speed | Change measure: Baseline, within one week after intervention, 6 weeks after intervention, 3 months after intervention, 6 months after intervention and 12 months after intervention
  40 meters Fast-Paced Walk test

SECONDARY OUTCOMES:
Change in physical function | Change measure: Baseline, within one week after intervention, 6 weeks after intervention, 3 months after intervention, 6 months after intervention and 12 months after intervention
  30 second sit-to stand test
Change in aerobic capacity | 1 week before intervention, directly after intervention as well as 6 and 12 weeks after TJA-surgery
  6 min walk test
Change in transitional ambulation | Change measure: Baseline, within one week after intervention, 6 weeks after intervention, 3 months after intervention, 6 months after intervention and 12 months after intervention
  Timed-up and go Test (TUG)
Change in pain measured with numeric rating scale (NRS) | Change measure: Baseline, within one week after intervention, 6 weeks after intervention and 3 months after intervention
  NRS - Single score, low score indicates low pain, high score indicated high levels of pain
Length of stay in hospital | From date of hospital admission until the date of hospital discharge, assessed up to 12 months
  Number of days
Change in the ability to climb stairs | Change measure: Baseline, within one week after intervention, 6 weeks after intervention, 3 months after intervention, 6 months after intervention and 12 months after intervention
  Stair-climb test. Timed performance from start to stop
Change in Health Status measured with EuroQol-5 dimensions (EQ-5D) | Change measure: Baseline, within one week after intervention, 6 weeks after intervention, 3 months after intervention, 6 months after intervention and 12 months after intervention
  EQ-5D, five dimensions of health scored from 1-5, with 1 being no problem and 2-5 indicate increasing problem (higher score = increase in problem)

CONTACTS AND LOCATIONS:
Overall Officials: Odd-Einar Svinøy, MSc, Principal Investigator — OsloMet
Locations (1):
- OsloMet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Slatkowsky-Christensen B, Grotle M. Artrose i Norge. Norsk Epidemiologi 2008;18(1)
- [Background] Wallace IJ, Worthington S, Felson DT, Jurmain RD, Wren KT, Maijanen H, Woods RJ, Lieberman DE. Knee osteoarthritis has doubled in prevalence since the mid-20th century. Proc Natl Acad Sci U S A. 2017 Aug 29;114(35):9332-9336. doi: 10.1073/pnas.1703856114. Epub 2017 Aug 14. PMID 28808025
- [Background] Bitton R. The economic burden of osteoarthritis. Am J Manag Care. 2009 Sep;15(8 Suppl):S230-5. PMID 19817509
- [Derived] Svinoy OE, Nordbo JV, Pripp AH, Risberg MA, Bergland A, Borgen PO, Hilde G. The effect of prehabilitation for older patients awaiting total hip replacement. A randomized controlled trial with long-term follow up. BMC Musculoskelet Disord. 2025 Mar 6;26(1):227. doi: 10.1186/s12891-025-08468-4. PMID 40050814
- [Derived] Svinoy OE, Bergland A, Risberg MA, Pripp AH, Hilde G. Better before-better after: efficacy of prehabilitation for older patients with osteoarthritis awaiting total hip replacement-a study protocol for a randomised controlled trial in South-Eastern Norway. BMJ Open. 2019 Dec 30;9(12):e031626. doi: 10.1136/bmjopen-2019-031626. PMID 31892650